CLINICAL TRIAL: NCT02574169
Title: Alveolar Recruitment Maneuvers, Intracerebral Hemodynamic and Oxygenation
Acronym: M'RHICO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RC31/15/7604
Record Dates: First submitted 2015-09-19; First posted 2015-10-12 (Estimated); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Cerebral Injuries; Acute Respiratory Distress Syndrome (ARDS)
Keywords: Alveolar Recruitment Maneuvers (ARM); Continuous Positive Airway Pressure (CPAP); Extended Sigh (eSigh)
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alveolar recruitment maneuvers Group 1 (Experimental): alveolar recruitment maneuvers by CPAP then alveolar recruitment maneuvers by eSigh
  Interventions: Other: alveolar recruitment maneuvers group 1
- Alveolar recruitment maneuvers Group 2 (Experimental): alveolar recruitment maneuvers by eSigh then alveolar recruitment maneuvers by CPAP
  Interventions: Other: alveolar recruitment maneuvers group 2

INTERVENTIONS:
Other: alveolar recruitment maneuvers group 1 — Patients are randomized to receive in cross-over 2 ARM: CPAP at first and then eSigh.
  The continuous positive airway pressure, or CPAP with application of a positive pressure of 40 cmH2O for 40 seconds without tidal volume.
  The eSigh or extended sigh with increase of PEEP for 10 minutes to maintain plateau pressure at 40 cmH2O. During ARM, the peak pressure is limited to 50 cmH2O with decrease of tidal volume (Vt) if necessary.
  The following data: PtiO2, respiratory parameters, systemic and intracerebral hemodynamic parameters are collected before, after 1 minute, 10 minutes and 60 minutes for each ARM.
  Arms: Alveolar recruitment maneuvers Group 1
Other: alveolar recruitment maneuvers group 2 — Patients are randomized to receive in cross-over 2 ARM: eSigh at first and then CPAP.
  The eSigh or extended sigh with increase of PEEP for 10 minutes to maintain plateau pressure at 40 cmH2O. During ARM, the peak pressure is limited to 50 cmH2O with decrease of tidal volume (Vt) if necessary.
  The continuous positive airway pressure, or CPAP with application of a positive pressure of 40 cmH2O for 40 seconds without tidal volume.
  The following data: PtiO2, respiratory parameters, systemic and intracerebral hemodynamic parameters are collected before, after 1 minute, 10 minutes and 60 minutes for each ARM.
  Arms: Alveolar recruitment maneuvers Group 2

SUMMARY:
This study aims to compare 2 alveolar recruitment maneuvers (ARM) in patients with cerebral injuries and acute respiratory distress syndrome (ARDS) in term of efficacy and tolerance.

DETAILED DESCRIPTION:
Two ARM are compared in this study:

* The eSigh or extended sigh with increase of PEEP for 10 minutes to maintain plateau pressure at 40 cmH2O. During ARM, the peak pressure is limited to 50 cm H2O with decrease of tidal volume (Vt) if necessary.
* The continuous positive airway pressure, or Continuous Positive Airway Pressure (CPAP) with application of a positive pressure of 40 cm H2O for 40 seconds without tidal volume.

Patients are randomized to receive in cross-over 2 ARM: CPAP and Extended Sigh (eSigh). The following data: oxygen tissue partial pressure (PtiO2), respiratory parameters, systemic and intracerebral hemodynamic parameters are collected before, after 1 minute, 10 minutes and 60 minutes for each ARM.

ELIGIBILITY:
Inclusion Criteria:

* Patients with brain injuries (subarachnoid hemorrhage, traumatic brain injury, ischemic and hemorrhagic stroke)
* Patients with moderate and severe ARDS criteria (as defined by classification of Berlin)
* Patients under mechanical ventilation

Exclusion Criteria:

* ICP (Intracranial pressure) > 25 mmHg
* Pregnant women
* Patients with history of chronic respiratory disease
* Patients with bronchopleural fistula
* Patients with hemodynamic instability despite appropriate measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of oxygen tissue partial pressure (PtiO2) values | 60 minutes
  The comparison of PtiO2 values (mmHg, mean ± SD) 60 minutes after the 2 ARM: eSigh and CPAP

SECONDARY OUTCOMES:
Comparison of systemic hemodynamic parameters | 60 minutes
  Comparison between the two ARM of systemic hemodynamic parameters: mean arterial pressure, heart rate and cardiac output.
Comparison of Intracranial hemodynamic parameters | 60 minutes
  Comparison between the two ARM of Intracranial hemodynamic parameters: ICP (Intracranial pressure) , cerebral perfusion pressure and Transcranial Doppler (pulsatility index, mean, systolic and diastolic velocities)
Comparison of blood oxygen level | 60 minutes
  Comparison between the two ARM of haematosis: Blood oxygen level (SpO2)
Comparison of partial pressure of carbon dioxide | 60 minutes
  Comparison between the two ARM of partial pressure of carbon dioxide (PaCO2),
Comparison of arterial blood gases | 60 minutes
  Comparison between the two ARM of arterial blood gases (partial pressure of oxygen (PaO2),
Comparison of end-tidal CO2 | 60 minutes
  Comparison between the two ARM of end-tidal CO2
Comparison of Respiratory parameters | 60 minutes
  Comparison between the two ARM of Respiratory parameters: plateau pressure and static lung compliance.
Comparison of PtiO2 | 60 minutes
  Comparison between the two ARM of PtiO2

CONTACTS AND LOCATIONS:
Overall Officials: Ségolène MROZEK, MD, Principal Investigator — UH TOULOUSE
Locations (5):
- France (5):
  - UH Toulouse, Toulouse, Midi Pyrénées
  - UH Caen, Caen
  - UH Clermont-Ferrand, Clermont-Ferrand
  - UH Montpellier, Montpellier
  - UH Nantes, Nantes

REFERENCES:
- [Background] Constantin JM, Jaber S, Futier E, Cayot-Constantin S, Verny-Pic M, Jung B, Bailly A, Guerin R, Bazin JE. Respiratory effects of different recruitment maneuvers in acute respiratory distress syndrome. Crit Care. 2008;12(2):R50. doi: 10.1186/cc6869. Epub 2008 Apr 16. PMID 18416847
- [Background] Rangel-Castilla L, Gopinath S, Robertson CS. Management of intracranial hypertension. Neurol Clin. 2008 May;26(2):521-41, x. doi: 10.1016/j.ncl.2008.02.003. PMID 18514825
- [Background] Chesnut RM. Care of central nervous system injuries. Surg Clin North Am. 2007 Feb;87(1):119-56, vii. doi: 10.1016/j.suc.2006.09.018. PMID 17127126
- [Background] Briel M, Meade M, Mercat A, Brower RG, Talmor D, Walter SD, Slutsky AS, Pullenayegum E, Zhou Q, Cook D, Brochard L, Richard JC, Lamontagne F, Bhatnagar N, Stewart TE, Guyatt G. Higher vs lower positive end-expiratory pressure in patients with acute lung injury and acute respiratory distress syndrome: systematic review and meta-analysis. JAMA. 2010 Mar 3;303(9):865-73. doi: 10.1001/jama.2010.218. PMID 20197533